CLINICAL TRIAL: NCT02216032
Title: Thirty Million Words Home Visiting: A Longitudinal RCT
Brief Title: Thirty Million Words Home Visiting
Acronym: TMW HV RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14-0895
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Language Environments of Children of Low-socioeconomic Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): We will deliver the TMW Curriculum to 106 Treatment families. The TMW Curriculum is comprised of 1) 12 educational modules, 2) animations and videos of real parent-child interactions to teach parents about the science behind child brain development, and model strategies for improving parents' child-directed speech, 3) video modeling and collaborative goal setting, and 4) quantitative linguistic feedback from Language ENvironment Analysis (LENA) recordings.
  Interventions: Other: TMW Curriculum
- Control Group (Other): We will deliver a Nutrition Curriculum to 100 Control families. The Nutrition Curriculum provides information about the importance of healthy nutrition for child development, strategies for healthy eating, and meal preparation.
  Interventions: Other: Nutrition Curriculum

INTERVENTIONS:
Other: TMW Curriculum
  Arms: Treatment Group
Other: Nutrition Curriculum
  Arms: Control Group

SUMMARY:
The TMW intervention aims to foster parental behaviors that facilitate children's language emergence at a critical developmental stage, and thus will be implemented at 13-16 months of age. The investigators hypothesize that the primary effects of the TMW Intervention will significantly 1) improve low-SES parents' understanding of the importance of parent language in a child's development, 2) increase parents' linguistic interaction, responsiveness, and overall engagement with their children, and 3) increase children's language output, as measured through LENA (child vocalization count, conversational turn count), coded video interaction (number of types, tokens and utterances for both children and adults), audio recordings from The Three T's application during the video sessions, and a battery of assessments targeting linguistic and cognitive development. Furthermore, the investigators hypothesize that increased parental interaction will result in 4) an improvement in children's socioemotional development as assessed by the Social Emotional Ages and Stages Questionnaire (ASQ-SE). Finally, the investigators hypothesize that these socioemotional and linguistic gains through early development, along with sustained increased parental engagement, will be expressed in 5) increased child school readiness upon kindergarten entry as assessed by Woodcock-Johnson Psycho-Educational Battery (WJ).

Added 2023: an 8th child-assessment, parent/child interaction video session, and parent surveys have been added with the original sample to measure long-term outcomes of children whose parents participated in the home visiting intervention.

DETAILED DESCRIPTION:
During the Recruitment Phase, a TMW research assistant (RA) will recruit participants for the study. If interested in joining the study, participants will complete the Preliminary Enrollment Consent. From this point forward, all study activities will take place in the participant's home. To follow the completion of the Preliminary Enrollment Consent, participants will be asked to complete a series of baseline measurements over a four-week time period. RAs will facilitate the collection of these measures. Following satisfactory completion of the baseline measures, participants will move on to the Enrollment Phase at which point they will complete the Enrollment Consent. At this point, participants will be randomized into either one of two conditions (The Treatment group received an educational curriculum on language development and the Control group receives an educational curriculum on the role of nutrition in development) as part of a matched pair. Pairs will be matched by 1) age of the child and 2) averaged conversational turn counts from the 3 baseline LENA recordings. Assignment to Control or Treatment of each member of a pair is decided through a coin flip. Additionally, participants will complete Video 1, administered by an RA. During this and all subsequent Videos, audio recordings will be taken using both the LENA and the Three T's App. Following the Enrollment Phase, participants will move on to the Intervention Phase. During the Intervention Phase, participants will first complete Assessment 1. A staff member of Thirty Million Words will conduct this and all subsequent assessments. Following Assessment 1, participants will receive 12 bi-weekly home visits over a six-month period from trained TMW Home Visitors. During the home visits, Home Visitors will deliver two different curricula to the respective groups. The Treatment group will receive the TMW Curriculum. The Control group will receive the alternative Nutrition Curriculum, which provides information about the importance of healthy nutrition for child development, strategies for healthy eating, and meal preparation. In addition to receiving the home visits, participants will also complete LENA recordings on a bi-weekly basis, alternating weeks with the home visiting schedule. Participants in both the Control and the Treatment condition will receive text messages to remind them to complete their LENA recording on the day that they had previously scheduled. For the Treatment group only, a text message reminder for a specific goal will be sent as well. This will help parents be mindful of their goals at the time that they plan to achieve them by reminding parents to engage linguistically with their children. This text reminder portion of the study will piggy-back on the goal setting portions in which the parent will set specific, personalized goals. Reminders of these goals will be sent to their phones at a day and time that parents choose. Both the Treatment and Control participants will be given the option to opt out of the text messaging if they do not wish to receive these messages. Following the Intervention Phase, participants will move on to the 42-month Follow-up Phase. Throughout this phase, participants will complete Videos 2-7 with an RA, Assessments 2-7 with a TMW assessor, LENA recordings 16-21, and four curricula supplementation 'Boosters,' delivered by an RA. This marks the final phase of involving participants. After study completion, Dr. Suskind or her research team will contact participants regarding theirs and their child's participation in further research studies. A separate IRB protocol will be submitted at that time.

Transcription Service Feasibility Pilot Study

The purpose of this pilot study is to assess the feasibility of using a transcription service to transcribe Video Session recordings compared to using University of Chicago research personnel. Up to 10 already enrolled participants will be asked to participate in a pilot study to assess the feasibility of using a transcription service to transcribe participant Video Session recordings. Each participant in the pilot study will receive an addendum to the study consent document and discuss the addendum with a member of the research team prior to their study video sessions being sent to third-party transcription services to conduct a feasibility study.

A Business Associate and Service Agreement is being processed between the University and the transcription service to ensure University approved security measures are in place to transcribe participant video sessions. No videos will be sent to the transcription service until the Business Associate and Service Agreement is approved.

Added 2023: when the children in the original sample turn 9-10 years old, parents are contacted with the opportunity to complete an additional study time point, to evaluate their child's outcomes as they've reached 3rd - 4th grade. Participants sign an addendum to the enrollment consent in order to participate. Trained assessors meet with the child to conduct measures of language, cognitive, and math skills ("Assessment 8"). Additionally, the assessor records a parent-child interaction completing an age-appropriate task ("Video Session 8"). Finally, the parent completes a series of surveys measuring knowledge about child development, parental inputs, and child behaviors

ELIGIBILITY:
Inclusion Criteria:

* participants (i.e. parents and their children) who live at or below 250% of the federal poverty line
* paternal education at or below BA/BS
* parents with children between the ages of 13-16 months old

Exclusion Criteria:

* participants (i.e. parents and their children) who live over 200% of the federal poverty line
* parents under the age of 18
* children younger than 13 months old or older than 16 months old (at start of study)
* parents who do not have legal custody of their child
* parents whose child does not live with them
* parents who are not with their child at least two full days per week
* parents who are unable to commit to the intervention requirements
* foster parents
* children with significant cognitive or physical impairments (specifically Autism Spectrum Disorder, Epilepsy, Cerebral Palsy, hearing impairment, Down Syndrome and blindness)
* parents who have earned or are currently working toward a graduate or professional degree (e.g. M.A., M.S., M.B.A)
* parents who speak less than 80% English to their children.

Ages: 13 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2014-11; Primary Completion 2022-01-16 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Preschool Language Scale IV (PLS) | Baseline, month 6, month 12, month 18, month 24, month 36, month 48
  The PLS is used as a measure of a child's receptive vocabulary, and is used in this study to evaluate a child's language development from baseline to Month 48. It is a direct to child assessment administered by a trained assessor. Raw score values range from 0 to 65, with a higher score indicating higher receptive vocabulary skills.
Peabody Picture Vocabulary Test (PPVT) | Month 24, Month 36, Month 48, Month 96
  The PPVT is a measure of a child's receptive vocabulary, and is used in this study to evaluate a child's language development from Month 24 to Month 48 and as a measure of school readiness upon kindergarten entry. It is additionally used to evaluate language development at Month 96. It is a direct to child assessment administered by a trained assessor. Raw score values range from 0 to 175, with a higher score indicating higher receptive vocabulary skills. It is a direct to child assessment administered by a trained assessor. This assessment is a primary outcome measure at Months 24, 36, and 48 and secondary at month 96.
Language ENvironment Analysis | Month 0, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 12, Month 18, Month 24, Month 36, Month 48
  LENA is a recording device that is worn by the child to provide metrics of conversational turn counts, adult word counts, and child vocalizations. LENA is used in this study as a quantitative measure of parent child interaction and to measure change from baseline in child oral language development and production to month 48.
Parent/Child video sessions | Month 0, Month 6, Month 12, Month 18, Month 24, Month 36, Month 48, Month 96.
  Observational coding is used to characterize quality of interactions between parent and child during recorded free-play and book sharing activities. This outcome is primary at months 0-48 and secondary at Month 96.

SECONDARY OUTCOMES:
Woodcock Johnson (WJ-IV). | Month 48, Month 96
  The WJ-IV is a measure of a child's achievement and cognitive abilities. It is used in this study as a measure of school readiness at kindergarten entry and skills in mid-elementary school. It is a direct to child assessment administered by a trained assessor. A higher score on this assessment indicates greater skills.
NIH toolbox Cognition Battery | Month 96
  The NIH toolbox Cognition Battery assesses a child's executive function skills, including inhibitory control and working memory. It is a direct to child assessment completed by the child using an iPad. A higher score on this assessment indicates greater executive function skills relative to other children of the same age. This additional outcome measure was added in 2023 with the addition of an 8th study assessment.
Ages and Stages Questionnaire: Social-Emotional (ASQ:SE) | Month 6, Month 24, Month 36, Month 48
  The ASQ:SE is a screening tool designed to capture concerns about a child's social-emotional development. It is a parent report measure used in this study as a measure of school readiness upon kindergarten entry. Score values range from 0 to 360, with a higher value indicating that a child's social-emotional development may not be at an age-appropriate level.
Give-a-number task (Give-N) | Month 36, Month 48
  The Give-N task is a measure of a child's understanding of number words. It is a direct to child assessment, administered by a trained assessor used in this study as a measure of school readiness upon kindergarten entry. Scores range from 0-6, with a higher score indicated that a child has a greater comprehension of number words.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Suskind, MD, Principal Investigator — University of Chicago
Locations (1):
- Thirty Million Words® Initiative at the University of Chicago Medicine, Chicago, Illinois, United States

REFERENCES:
- [Background] Suskind, D., Leffel, K. R., Hernandez, M. W., Sapolich, S. G., Suskind, E., Kirkham, E., & Meehan, P. (2013) An exploratory study of "Quantitative Linguistic Feedback": Effect of LENA Feedback on Adult Language Production. Communication Disorders Quarterly. 34(4) 199-209. Doi: 10.1177/1525740112473146
- [Derived] LoRe D, Leung CYY, Brenner L, Suskind DL. Parent-directed intervention in promoting knowledge of pediatric nutrition and healthy lifestyle among low-SES families with toddlers: A randomized controlled trial. Child Care Health Dev. 2019 Jul;45(4):518-522. doi: 10.1111/cch.12682. Epub 2019 May 27. PMID 31050026
- See also: Click here for more information about the Thirty Million Words — https://tmwcenter.uchicago.edu/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT02216032/Prot_SAP_004.pdf